CLINICAL TRIAL: NCT05964283
Title: Physician Knowledge Level of Intravenous Fluid Therapy in Hospitals: A Cross-Sectional Study
Brief Title: Intravenous Fluid Therapy in Hospitals
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal Investigator, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes047
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Knowledge Level; Intravenous Fluid Therapy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anesthesia Specialists
  Interventions: Other: Questionnaire
- Anesthesiologist residencies
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — This questionnaire consists of (five) main parts. The first part is about personal information, the second part is about fluid administration in various settings (emergency room, operating room, and intensive care unit), the third part is about fluid administration behaviors, the fourth part is about workplace location, and the fifth part is about a case study. Filling out this questionnaire will take approximately 60 minutes of your time.

SUMMARY:
The administration of intravenous fluids plays a crucial role in critically ill patients to support optimal management and ensure patient safety. Knowledge and conceptual frameworks will influence a clinician's accuracy in providing intravenous fluid therapy to patients. Accurate administration of fluid therapy to patients will reduce unwanted side effects and decrease the overall treatment costs during hospitalization. Various considerations in administering intravenous fluid therapy are influenced by a clinician's level of knowledge. In Indonesia, doctors working in hospitals may have different levels of education and professional status. However, it is currently unclear whether these professional differences among doctors influence their knowledge in administering fluids to patients.

ELIGIBILITY:
Inclusion Criteria:

* All anesthesiologist residencies and are willing to complete the questionnaire.
* All anesthesia specialists and subspecialists and are willing to complete the questionnaire until finished.

Exclusion Criteria:

* All doctors who are unwilling and do not complete the survey questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Anesthesia specialists
  * Anesthesiologist residencies
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire regarding Physician Knowledge Level of Intravenous fluid therapy | one day
  Intravenous Fluid Therapy knowledge Scoring
  The principle for scoring these scales is the same in all cases:
  1. Estimate the average of the items that contribute to the scale; this is the raw score. Calculating the raw score=(I1+I2+I3+…+In)/n.
  2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of knowledge. Formula use for standardization: Knowledge Score = {1-(Raw score-1)/range} X100
  The maximum score is 100 (better outcome) The minimum score is 0 (worse outcome)
  All the information related to intravenous fluid therapy is divided into five domains: (1) basic knowledge about electrolyte fluids, (2) intravenous fluid administration, (3) intravenous fluid composition, (4) fluid resuscitation, and (5) assessment of fluid volume status.

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, Principal Investigator — Indonesia University
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malbrain MLNG, Langer T, Annane D, Gattinoni L, Elbers P, Hahn RG, De Laet I, Minini A, Wong A, Ince C, Muckart D, Mythen M, Caironi P, Van Regenmortel N. Intravenous fluid therapy in the perioperative and critical care setting: Executive summary of the International Fluid Academy (IFA). Ann Intensive Care. 2020 May 24;10(1):64. doi: 10.1186/s13613-020-00679-3. PMID 32449147
- [Background] McDougall M, Guthrie B, Doyle A, Timmins A, Bateson M, Ridley E, Drummond G, Vadiveloo T. Introducing NICE guidelines for intravenous fluid therapy into a district general hospital. BMJ Open Qual. 2022 Feb;11(1):e001636. doi: 10.1136/bmjoq-2021-001636. PMID 35115322
- [Background] Finfer S, Myburgh J, Bellomo R. Intravenous fluid therapy in critically ill adults. Nat Rev Nephrol. 2018 Sep;14(9):541-557. doi: 10.1038/s41581-018-0044-0. PMID 30072710
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Tommasino C. Fluids and the neurosurgical patient. Anesthesiol Clin North Am. 2002 Jun;20(2):329-46, vi. doi: 10.1016/s0889-8537(01)00013-x. PMID 12165997
- [Background] Rudloff E, Hopper K. Crystalloid and Colloid Compositions and Their Impact. Front Vet Sci. 2021 Mar 31;8:639848. doi: 10.3389/fvets.2021.639848. eCollection 2021. PMID 33869319
- [Background] Mackenzie DC, Noble VE. Assessing volume status and fluid responsiveness in the emergency department. Clin Exp Emerg Med. 2014 Dec 31;1(2):67-77. doi: 10.15441/ceem.14.040. eCollection 2014 Dec. PMID 27752556